CLINICAL TRIAL: NCT02847585
Title: Potential Role of Water-soluble Ubiquinol in Complementary Therapy for Pediatric Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yeh, Principal Investigator, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MOST105-2628-B-040-MY2
Record Dates: First submitted 2016-07-12; First posted 2016-07-28 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Dilated Cardiomyopathy
Keywords: water-soluble ubiquinol supplementation; pediatric cardiomyopathy; antioxidant; inflammation; complementary therapy
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): water-soluble ubiquinol
  Interventions: Dietary Supplement: Water-soluble Ubiquinol

INTERVENTIONS:
Dietary Supplement: Water-soluble Ubiquinol — 10 mg/kg BW/d, by oral drops

SUMMARY:
Pediatric dilated cardiomyopathy (PDCM) is the most common form fond in children. Water-soluble coenzyme Q10 (ubiquinol) is better absorbed than lipid-soluble coenzyme Q10 (ubiquinone) and is directly involved in the antioxidant cycle. Because coenzyme Q10 has shown significant health benefits in adult patients with cardiovascular disease, it is worth studying water-soluble coenzyme Q10 supplements to evaluate their potential role as complementary therapy for PDCM. The purpose of this study is to explore the potential role of water-soluble ubiquinol in complementary therapy for pediatric cardiomyopathy. We will recruit 25 children with primary PDCM (age 0-20 y) and examine the relationship between coenzyme Q10 level and cardiac function (left ventricular fractional shortening and ejection fraction, and B-type natriuretic peptide), oxidative stress (malondialdehyde), antioxidant enzymes activity (catalase, glutathione peroxide, and superoxide dismutase), and inflammation (high sensitivity C-reactive protein and interleukin-6) in PMC after 6 months water-soluble ubiquinol supplementation (10 mg/kg BW/d, by oral drops). In addition, we will assess the quality of life of PDCM patients by questionnaire. Through this study, we expect to demonstrate that water-soluble coenzyme Q10 will be a complementary therapy for PDCM, and will improve cardiac function, increase antioxidant capacity, slow deterioration of cardiac function and reduce inflammation, and further reduce the rate of heart transplantation and increase quality of life in PDCM.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric dilated cardiomyopathy defined as left ventricular ejection fraction ≤ 40 % by cardiac echo examination.

Exclusion Criteria:

* Hypertension
* Arrhythmia
* Congenital heart defects
* Acute myocarditis
* Pregnant and lactating teens
* Antioxidant vitamins users

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 6 months
  Left ventricular ejection fraction (%) will be measured by cardiac echo.

SECONDARY OUTCOMES:
Levels of plasma coenzyme Q10 | 6 months
  Plasma coenzyme Q10 (micromol/L) will be measured by high performance liquid chromatography.
B-type natriuretic peptide (BNP) | 6 months
  BNP (pg/mL) will be measured by fluorescence immunoassay.
malondialdehyde (MDA) | 6 months
  MDA (micromol/L) will be measured by thiobarbituric acid reacting substance.
catalase (CAT) | 6 months
  red blood cells level of CAT in unit/mg protein.
glutathione peroxide (GPx) | 6 months
  red blood cells level of GPx in unit/mg protein.
superoxide dismutase (SOD) | 6 months
  red blood cells level of SOD in unit/mg protein.
high sensitivity C-reactive protein (hs-CRP) | 6 months
  hs-CRP (mg/dL) will be measured by Immunoturbidimetry.
high sensitivity interleukin-6 (IL-6) | 6 months
  IL-6 (pg/dL) will be measured by immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ting Lin, Ph.D., Principal Investigator — School of Nutrition, Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No